CLINICAL TRIAL: NCT07091084
Title: Herbal Formula Ma-Zi-Ren-Wan (MZRW) on Bowel Movement Function and Gut Microbiome Among Cancer Survivors With Constipation: A Double-blinded Randomized Controlled Trial (RELIEVE)
Brief Title: A Study of Herbal Supplements in Cancer Survivors With Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-076
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Constipation; Cancer; Functional Constipation
Keywords: constipation; functional constipation; Ma-Zi-Ren-Wan; MZRW; 25-076; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Constipation; Neoplasms | interventions — ma zi ren wan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MZRW (Experimental): Participants will receive 2 weeks of MZRW
  Interventions: Dietary Supplement: MZRW
- Placebo (No Intervention): Participants will receive 2 weeks of placebo

INTERVENTIONS:
Dietary Supplement: MZRW — MZRW herbal formula consists of a 7:1 extract of Huo Ma Ren [Hemp Seed 33.4%]; Da Huang (Sheng) [Rhubarb (Fresh) 22.2%]; Bai Shao [Peony (White) 11.1%]; Zhi Shi [Aurantium Immaturus 11.1%]; Hou Po [Magnolia Bark 11.1%]; and Xing Ren [Apricot Kernel 11.1%] - Taken for 2 weeks intervention and 2 weeks follow-up
  Other Names: Ma-Zi-Ren-Wan
  Arms: MZRW

SUMMARY:
The purpose of this study is to find out whether MZRW is an effective treatment for constipation in cancer survivors. The researchers will compare MZRW with placebo, a pill that looks like MZRW and is given in the same way, but contains no medication. The researchers will also study the effect MZRW has on the gut microbiome. The gut microbiome is a diverse community of microorganisms living in the digestive system, essential for digestion and immune function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater;
* A diagnosis of cancer with no restrictions placed on type of cancer or stage;
* Completed surgery, chemotherapy, immunotherapy, and/or radiotherapy, or an investigational therapy at least one month prior to study initiation. Patients on stable doses of hormone therapy or targeted therapies will not be excluded;
* Karnofsky functional score of ≥ 60;
* Cancer survivors who have met the Rome IV criteria (Table 3) of the symptoms of functional constipation which must include two or more of the following:

  * Straining more than 25% of defecations.
  * Lumpy or hard stools (7-point Bristol stool scale 1 or 2) more than 25% of defecations.
  * Sensation of incomplete evacuation more than one-fourth (25%) of defecations.
  * Sensation of anorectal obstruction/blockage more than one-fourth (25%) of defecations.
  * Manual maneuvers to facilitate more than one-fourth (25%) of defecations.
  * Fewer than three spontaneous bowel movements per week.
  * Loose stools are rarely present without the use of laxatives.
  * Insufficient criteria for irritable bowel syndrome.
* Patient should be able to understand and complete all study assessments on their own
* Patient should be able to understand and provide signed informed consent in English.

Table 3. Rome IV criteria for functional constipation FUNCTIONAL CONSTIPATION Diagnostic criteria*

1. Must include two or more of the following:**
2. Straining during more than ¼ (25%) of defecations
3. Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations
4. Sensation of incomplete evacuation more than ¼ (25%) of defecations
5. Sensation of anorectal obstruction/blockage more than ¼ (25%) of defecations
6. Fewer than three SBM per week
7. Manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor)

9. Loose stools are rarely present without the use of laxatives 9. Insufficient criteria for irritable bowel syndrome Note *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis

Exclusion Criteria:

* Patients who have allergic history to herbs or Chinese medicine;
* Clinically significant abnormal liver (2 times the ULN for ALT or AST) and kidney disfunction(eGFR below 59 mL/min/1.73m² ) from recent laboratory test recorded in the medical record (within 1 month);
* Patients who have any signs of bowel obstruction, or have high risk of bowel obstruction assessed by their treating physician, including factors such as tumor invasion into abdominal organs, recent abdominal surgery, and prior abdominal radiation therapy;
* Patients who are prescribed opioid antagonists including methylnaltrexone, naloxegol and naldemedine for opioid induced constipation and required not to stop the medication;
* Women who are pregnant, lactating, or not practicing proper contraception by patient report.Patient's should follow proper contraception guidelines for at least 30 days following last dose of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Difference of spontaneous bowel movements (SBMs) from baseline to week 2 | 2 weeks
  To evaluate the efficacy of a 2-week regimen of oral MZRW vs. placebo on spontaneous bowel movements (SBMs), in terms of SBM therapeutic response (primary efficacy endpoint), among cancer survivors with chronic constipation. SBM response is defined at week 2 as having an increase of ≥ 1 SBM/week from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org